CLINICAL TRIAL: NCT04672967
Title: Metabolic Autism Prediction (MAP) Study
Brief Title: MAP Autism Prediction Study
Acronym: MAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BioROSA Technologies Inc (Industry)
Collaborators: Melmed Center (Unknown); Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: 1320036
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Autism Spectrum Disorder; Developmental Delay
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fasting plasma samples will be collected to evaluate metabolites and other biomarkers which may be predictive of ASD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder: Children diagnosed with ASD between the ages of 18-60 months
  Interventions: Diagnostic Test: BioROSA MAP test
- Non-ASD (developmental delay or typically developing): Children diagnosed with non-ASD between the ages of 18-60 months
  Interventions: Diagnostic Test: BioROSA MAP test

INTERVENTIONS:
Diagnostic Test: BioROSA MAP test — The BioROSA MAP test is a blood test that is being developed to predict ASD risk

SUMMARY:
This pilot clinical trial tests the hypothesis that certain blood metabolite levels can be used to predict Autism Spectrum Disorder (ASD). The study cohort will consist of 200 participants between the ages 18 and 60 months who have been referred to a developmental pediatric center for clinical evaluation of ASD or other developmental delay. Two selected sites will enroll 75 participants each with another 50 typically developing participants. Participants will receive a physical exam (including a dysmorphology evaluation), ADOS, VABS, MSEL, DSM-5, and M-CHAT assessments, and receive a diagnosis. A fasting blood draw is required, consisting of 2 mL vacutainer tubes (max 4 mL). Sites must process blood according to sponsor requirements (outlined in the Sponsor's Laboratory Manual). Certain metabolite levels in the blood will be used for diagnostic screening test development.

DETAILED DESCRIPTION:
The primary objective is to conduct a double-blind, proof-of-concept, two-site, prospective study of 200 children aged 18-60 months that have been referred for an ASD evaluation by a physician to assess the feasibility of a blood test that measures a set of blood plasma metabolites and the classification algorithm developed thereof to predict the risk of ASD.

The secondary objective is to collect additional information for sub-classification of participant cohorts including Vineland Adaptive Behavior Scale (VABS) and Mullen Scale of Early Learning (MSEL) as well as any comorbidities that may correlate with blood test scores.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. 18-60 months of age
2. Primary language is English (this is due to the evaluation instruments being used, which are in the English language).
3. Suspected developmental concern and referral to the developmental center by child's physician
4. Parental informed consent to participate in the study (based on the age range of the children in this study, assent is being waived)
5. Willingness to comply with all study procedures
6. Not currently enrolled in another clinical trial

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Previous diagnosis of ASD or DD
2. Prematurity < 34 weeks' gestation
3. Has a sibling already enrolled in the trial
4. Profound sensory deficits (e.g., hearing and vision deficits) that could interfere with the interpretation of study results
5. Documented current or active seizures, as defined by a clinical seizure or abnormal EEG within the past six months
6. Major genetic defect as determined by chromosomal microarray or other method of genetic detection
7. Currently taking any high dose (greater than recommended daily allowance) dietary supplements
8. Diagnosis or suspicion of recent viral/bacterial infection within 2 weeks of enrollment
9. Diagnosis with congenital brain malformations, moderate to severe traumatic brain injury, congenital or acquired microcephaly, or infection of the central nervous system (e.g., meningitis, viral encephalitis)
10. Fetal alcohol syndrome, Down syndrome, or another recognized syndrome
11. Usage of acetaminophen (e.g., Tylenol) within the past 72 hours
12. Fever (temperature > 100 degrees Fahrenheit) within the past 72 hours
13. Any other reason that the clinical investigator feels may place the participant at an unnecessary risk to participate

Ages: 18 Months to 60 Months | Sex: All
Age Groups: Child
Study Population: Up to 250 participants, ages 18-60 months suspected of ASD or a developmental delay who are referred for evaluation at participating pediatric developmental centers.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Autism Diagnostic Observation Scale (ADOS) | 1 day (At study entry (one time evaluation))
  The Autism Diagnostic Observation Schedule (ADOS) is considered a gold-standard instrument for diagnosing and assessing autism with good diagnostic sensitivity and specificity in young children (37). The ADOS consists of a series of structured and semi-structured tasks that involve social interaction between the examiner and the person under assessment. The examiner observes and identifies segments of the subject's behavior and assigns these to predetermined observational categories. Categorized observations are subsequently combined to produce quantitative scores for analysis and diagnostic classification of ASD. Children at or above predetermined cutoff lines are considered to be positive for ASD.

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scale (VABS) | 1 day (At study entry (one time evaluation))
  Vineland Adaptive Behavior Scale (VABS). The Vineland Adaptive Behavior Scale (VABS) will measure functional abilities within several domains including communication, daily living skills, socialization, and motor skills. The VABS has been used widely in ASD assessments and provides a measure of core symptoms and adaptive function across a wide age range (38). All sections of the VABS up through physical activity "using small muscles" will be completed. Subsequent sections consisting of problem behaviors will not be completed, as these are not needed to obtain an adaptive behavior composite score.
Mullen Scales of Early Learning (MSEL) | 1 day (At study entry (one time evaluation))
  The Mullen Scales of Early Learning (MSEL) is a measure of cognitive functioning for infants and preschool-age children from birth through age 68 months. The MSEL is organized into 5 subscales: (a) gross motor, (b) fine motor, (c) visual reception (or non-verbal problem solving), (d) receptive language, and (e) expressive language. An early learning composite score can be derived from fine motor, visual reception, receptive language, and expressive language scales. For young children this early learning composite score is considered equivalent to a more traditional "IQ" score or a developmental standard score (38). Each subscale is standardized to calculate a standard score, percentile, and age-equivalent score.
Modiﬁed Checklist for Autism in Toddlers (M-CHAT) | 1 day (At study entry (one time evaluation))
  The M-CHAT is a 23 question (yes/no) parent-completed screening measure for ASD. The M-CHAT is a routinely used level 1 screening instrument for ASD and is recommended for universal screening for ASD at 18- and 24-month well baby visits by the American Academy of Pediatrics (AAP)

CONTACTS AND LOCATIONS:
Overall Officials: Raun Melmed, MD, Principal Investigator — Melmed Center
Locations (1):
- VUMC, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No